CLINICAL TRIAL: NCT05306457
Title: Human Neural Progenitor Cells Secreting Glial Cell Line-Derived Neurotrophic Factor (CNS10-NPC-GDNF) Delivered to the Motor Cortex for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: CNS10-NPC-GDNF Delivered to the Motor Cortex for ALS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Clive Svendsen, Executive Director, Board of Governors Regenerative Medicine Institute, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000278
Record Dates: First submitted 2021-12-21; First posted 2022-04-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Stem cells; Growth Factor; Regenerative; Neural Progenitor Cells; NPC; Transplantation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CNS10-NPC-GDNF - Group A (Experimental): Unilateral, Motor Cortex, 0.25x10^6 cells in 10 µL/site, 21 sites (5.25x10^6 total cells) - Motor cortex corresponding to the non-dominant hand
  Interventions: Biological: CNS10-NPC-GDNF
- CNS10-NPC-GDNF - Group B (Experimental): Unilateral, Motor Cortex, 0.5x10^6 cells in 10 µL/site, 21 sites (10.5x10^6 total cells) - Motor cortex corresponding to the non-dominant hand
  Interventions: Biological: CNS10-NPC-GDNF
- CNS10-NPC-GDNF - Group C (Experimental): Unilateral Motor Cortex, 0.5x10^6 cells in 10 µL/site, 21 sites (10.5x10^6 total cells) - Motor cortex corresponding to the dominant hand
  Interventions: Biological: CNS10-NPC-GDNF

INTERVENTIONS:
Biological: CNS10-NPC-GDNF — Unilateral injections of CNS10-NPC-GDNF into the motor cortex

SUMMARY:
The investigator is examining the safety of transplanting cells, that have been engineered to produce a growth factor, into the motor cortex (brain) of patients with Amyotrophic Lateral Sclerosis (ALS). The cells are called neural progenitor cells, which are a type of stem cell that can become several different types of cells in the nervous system. These cells have been derived to specifically become astrocytes, which is a type of neural cell. The growth factor is called glial cell line-derived neurotrophic factor, or GDNF. GDNF is a protein that promotes the survival of many types of neural cells. Therefore, the cells are called "CNS10-NPC-GDNF." The investigational treatment has been tested in people by delivering it to the spinal cord. However, it has only been delivered to the motor cortex of animals. In this study, we want to learn if CNS10-NPC-GDNF cells are safe to transplant into the motor cortex (brain) of people.

DETAILED DESCRIPTION:
This study will be the first to use a genetically modified progenitor cell line delivered to the motor cortex to treat a neurodegenerative disease. This is a Phase 1/2a, single-center, safety study of two escalating doses of human neural progenitor cells expressing GDNF (CNS10-NPC-GDNF) delivered unilaterally to the "hand-knob" area of the motor cortex of patients with ALS.

Subjects meeting all Eligibility Criteria and providing Informed Consent will be enrolled in one of three sequential dosing groups. Subjects will be treated sequentially with a minimum of one month interval between surgeries for the first three subjects in each dosing cohort. The remaining subjects in the cohort will be treated with a minimum interval of at least one week between surgeries.

Primary Outcome:

Safety, as evaluated by:

* Adverse Events and Serious Adverse Events
* Post-op MRI and/or CT (with contrast) and as clinically indicated

ELIGIBILITY:
Inclusion:

1. Confirmed diagnosis of ALS (Possible, Lab-supported Probable, Probable or Definite El Escorial Criteria)
2. Duration of ALS symptoms ≤ 36 months
3. Progressive weakness in upper extremities, with EMG supported evidence of denervation in both upper extremities
4. Forced Vital Capacity ≥50% of predicted normal in supine
5. Age: 18 years or older
6. Able to provide Informed Consent
7. Be geographically accessible to the study site and able to travel to study site for required visits
8. Have caregiver to assist in the transportation and care required by participation in the study
9. Not taking riluzole and/or edaravone or on a stable dose for ≥ 30 day
10. For women of child bearing capacity, negative pregnancy test prior to surgery and willingness to use birth control for the duration of the trial.
11. Medically able to undergo craniotomy as determined by the site PI and/or investigators
12. Medically able to tolerate the immunosuppression regimen as determined by the site PI

Exclusion:

1. Using invasive ventilatory assistance
2. Diagnosis of another active or unstable medical illness that may interfere with study participation at discretion of PI
3. Presence of any of the following conditions:

   1. Current drug or alcohol abuse
   2. Any known immunodeficiency syndrome
   3. Unstable medical condition
   4. Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening
4. Persons of child bearing capacity not willing to practice birth control
5. Receiving any investigational device/biologic/drug in the past 30 days or any previous exposure to stem cell therapy
6. Any condition in the upper extremities that precludes serial strength or coordination testing
7. Any condition that the investigators feel may pose complications for the surgery
8. Any condition or ALS disease phenotype that the site PI feels may interfere with participation in the study or in the interpretation of study endpoints
9. Allergy to Beta-Lactam antibiotics
10. Donor Specific Antibodies (DSA) ≥ 2500MFI or CPRA ≥ 20%
11. Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety, as evaluated by the incidence of Adverse Events and Serious Adverse Events and their relationship to the treatment | 12 months post-operatively
Safety, as evaluated by changes from baseline in the brain MRI | 12 months post-operatively

SECONDARY OUTCOMES:
Force Generation via Accurate Test of Limb Isometric Strength (ATLIS) testing | ATLIS testing will be performed 7 times over 15 months
  Change from baseline for force generation by ATLIS
Pinch Strength | Pinch Strength testing will be performed 7 times over 15 months
  Change from baseline for pinch strength
Hand/Wrist Strength | Hand/Wrist strength testing will be performed 7 times over 15 months
  Change from baseline for Hand/Wrist strength using Hand-held dynamometer
Compound Motor Action Potential (CMAP) | CMAP will be performed 7 times over 15 months
  Change from baseline for CMAP
Functional Hand assessments using 9-hole peg test | 9-hole peg testing will be performed 7 times over 15 months
  Change from baseline for 9-hole peg test
Penn Upper Motor Neuron Score (PUMNS) | PUMNS will be performed 7 times over 15 months
  Change from baseline for Penn Upper Motor Neuron Score. (Scale of 0-32, where 0 is normal)
Hand Knob - Functional MRI (fMRI) | fMRI will be performed up to 4 times over 15 months
  Changes from baseline in brain activity in the hand knob area evaluated by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lewis, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No